CLINICAL TRIAL: NCT00789191
Title: Effect of Detemir and Sitagliptin on Blood Glucose Control in Subjects With Type 2 Diabetes Mellitus
Brief Title: Effect of Detemir and Sitagliptin on Blood Glucose Control in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-3511; 2008-001050-40 (EudraCT Number)
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Sitagliptin Phosphate; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comb (Experimental): Combination therapy of insulin detemir once daily plus sitagliptin added to subject's own pre-trial metformin treatment
  Interventions: Drug: insulin detemir; Drug: sitagliptin; Drug: metformin
- Sita (Active Comparator): Monotherapy of sitagliptin once daily added to subject's own pre-trial metformin and/or sulphonylurea (SU) treatment
  Interventions: Drug: sitagliptin; Drug: metformin; Drug: sulphonylurea

INTERVENTIONS:
Drug: insulin detemir — The detemir insulin dose is injected subcutaneously (under the skin) once daily in the evening and will be titrated (individually adjusted) weekly throughout the trial.
  Arms: Comb
Drug: sitagliptin — The sitagliptin dose is 100 mg/ day and should be kept stable throughout the trial. Frequency of sitagliptin is once daily.
Drug: metformin — Metformin treatment with at least 1000 mg/ day. Dose and dosing frequency should remain unchanged throughout the trial.
Drug: sulphonylurea — Sulphonylurea (SU) dose and dosing frequency should initially remain unchanged. In case of hypoglycaemia SU dose may be reduced at the discretion of the investigator.
  Arms: Sita

SUMMARY:
This trial is conducted in Asia, Europe and North America. This trial aims for comparison of the effect on the glycemic control in subjects with type 2 diabetes of basal insulin analogue with one oral anti-diabetic drug (OAD) versus oral anti-diabetic drug alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for at least 6 months before trial start
* Treatment with at least 1000 mg metformin per day for at least 3 months
* Insulin-naive (short-term insulin treatment of up to 14 days is allowed)
* DPP-4 (dipeptidyl peptidase-4) inhibitor naive
* HbA1c (glycosylated haemoglobin A1c) between 7.5-10.0% by central laboratory analysis
* BMI (Body Mass Index) lesser than or equal to 45.0 kg/m2
* Able and willing to take one subcutaneous injection every day
* Able and willing to perform mandatory SMPG (self measured plasma glucose) measurements

Exclusion Criteria:

* Known or suspected allergy or intolerance to any of the trial products or related products
* Severe hypertension
* Treatment with thiazolidinedione (TZD) or GLP-1 (glucagon-like peptide-1) analogues within 2 months prior to trial start
* Cardiac disease, within the last 12 months
* Impaired hepatic function
* Impaired renal function
* Proliferative retinopathy or macular oedema requiring acute treatment
* Female of childbearing potential
* Known or suspected abuse of alcohol, narcotics or illicit substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (46):
- United States (10):
  - Novo Nordisk Investigational Site, Vestavia Hills, Alabama
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Santa Monica, California
  - Novo Nordisk Investigational Site, Dunwoody, Georgia
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
- Canada (9):
  - Novo Nordisk Investigational Site, Coquitlam, British Columbia
  - Novo Nordisk Investigational Site, New Westminster, British Columbia
  - Novo Nordisk Investigational Site, St. John's, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Cambridge, Ontario
  - Novo Nordisk Investigational Site, Niagara Falls, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Saint Romuald, Quebec
  - Novo Nordisk Investigational Site, Sherbrooke, Quebec
  - Novo Nordisk Investigational Site, Niagara Falls
- Finland (6):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Loimaa
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Pieksämäki
  - Novo Nordisk Investigational Site, Pori
  - Novo Nordisk Investigational Site, Seinäjoki
- France (7):
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, La Roche-sur-Yon
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Montigny-lès-Metz
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Roubaix
- Hungary (3):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Eger
  - Novo Nordisk Investigational Site, Pécs
- Slovakia (5):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Lučenec
  - Novo Nordisk Investigational Site, Prešov
  - Novo Nordisk Investigational Site, Žilina
- South Korea (3):
  - Novo Nordisk Investigational Site, Daegu
  - Novo Nordisk Investigational Site, Incheon
  - Novo Nordisk Investigational Site, Seoul
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Kocaeli

REFERENCES:
- [Result] Hollander P, Raslova K, Skjoth TV, Rastam J, Liutkus JF. Efficacy and safety of insulin detemir once daily in combination with sitagliptin and metformin: the TRANSITION randomized controlled trial. Diabetes Obes Metab. 2011 Mar;13(3):268-75. doi: 10.1111/j.1463-1326.2010.01351.x. PMID 21205123
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 48 sites in 8 countries: Canada, Finland, France, Hungary, Slovakia, Republic of Korea, Turkey, and the United States of America (USA)
Pre-assignment Details: Between screening and randomisation, eligible subjects were to continue their usual pre-trial oral anti-diabetic drug (OAD) dose and dosing frequency. Subjects on sulphonylurea (SU) treatment randomised to the insulin detemir group had their SU discontinued
Period: Overall Study
Arm/Group | Comb | Sita
Started | 111 | 111
Exposed | 107 (2 withdrew informed consent. 1 randomised by mistake. 1 non-compliance) | 110 (1 non-compliance)
Completed | 97 | 92
Not Completed | 14 | 19
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 0 | 5
Not completed — Protocol Violation | 5 | 3
Not completed — Withdrawal Criteria | 2 | 4
Not completed — Unclassified | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Comb | Sita | Total
Number analyzed (Participants) | 107 | 110 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.70 (9.96) | 57.10 (8.41) | 56.90 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 60 | 99
  Male | 68 | 50 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 96 | 101 | 197
  Unknown or Not Reported | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 17 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 83 | 84 | 167
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 15
HbA1c [Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin] — HbA1c = glycosylated haemoglobin A1c
  Percent (%) glycosylated haemoglobin | 8.52 (0.65) | 8.52 (0.65) | 8.52 (0.65)
Height [Mean (Standard Deviation); unit: meters] | 1.71 (0.10) | 1.66 (0.09) | 1.68 (0.10)
Body Weight [Mean (Standard Deviation); unit: kg] | 93.1 (20.2) | 88.2 (19.2) | 90.6 (19.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI = Body Mass Index
  kg/m^2 | 31.79 (5.20) | 31.90 (5.91) | 31.85 (5.56)
Stratification [Number; unit: participants] — Previous OAD treatment
  participants
    Previous Metformin + Other OAD therapy | 83 | 86 | 169
    Previous Metformin Monotherapy | 24 | 24 | 48
FPG [Mean (Standard Deviation); unit: mmol/L] — FPG = Fasting Plasma Glucose
  mmol/L | 9.69 (2.23) | 9.79 (2.36) | 9.74 (2.29)
Diabetes History [Mean (Standard Deviation); unit: years] — No. of years subject has been diagnosed with diabetes
  years | 9.58 (5.62) | 9.90 (5.65) | 9.74 (5.63)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c (Glycosylated Haemoglobin A1c)
Time Frame: Week 26
Population: Sample size calculation: Assuming a standard deviation of 1.0 for HbA1c, 100 subjects in each treatment arm would be required to obtain a power of 80% for detecting a HbA1c difference of 0.4%. FAS (Full Analysis Set) is all randomised subjects exposed to at least one dose of trial product with a post baseline observation.
Measure: Mean (Standard Error); unit: Percent (%) glycosylated haemoglobin
Arm/Group | Comb | Sita
Number analyzed (Participants) | 103 | 106
Percent (%) glycosylated haemoglobin | 7.08 (0.09) | 7.64 (0.09)
Statistical Analysis 1: Comparison: Comb vs Sita; Null hypothesis: Difference between mean HbA1c in the two treatment arms is equal to zero. Power calculation: Assuming a standard deviation of 1.0 for HbA1c, 100 subjects in each treatment arm would be required to obtain a power of 80% for detecting a HbA1c difference of 0.4%; Test type: Superiority or Other; p = 0.0010, ANCOVA — No corrections to adjust for multiplicity were performed. Statistical significance threshold was p<0.05; Analysis of covariance (ANCOVA) was used; baseline HbA1c was included as covariate and treatment, stratification and country was included as factors; Mean Difference (Final Values) = -0.55, 95% CI [-0.77 to -0.33]

2. Secondary Outcome: Number of Subjects Achieving HbA1c Less Than or Equal to 7.0%
Time Frame: Week 26
Population: FAS (Full Analysis Set) is all randomised subjects exposed to at least one dose of trial product with a post baseline observation.
Measure: Number; unit: Subjects
Arm/Group | Comb | Sita
Number analyzed (Participants) | 103 | 106
Subjects
  Target achieved | 46 | 25
  Target not achieved | 57 | 81
Statistical Analysis 1: Comparison: Comb vs Sita; Null hypothesis: Odds ratio is equal to one; Test type: Superiority or Other; p = 0.0010, Regression, Logistic — No corrections to adjust for multiplicity were performed. Statistical significance threshold was p<0.05; Treatment group comparison using logistic regression model incl.treatment,stratification factor, country as fixed effects, baseline HbA1c as covariate; Odds Ratio (OR) = 3.20, 95% CI [1.65 to 6.19]

3. Secondary Outcome: Number of Subjects Achieving HbA1c Less Than or Equal to 7.0% Without Symptomatic Hypoglycaemia
Description: Symptomatic hypoglycaemia is biochemically confirmed hypoglycaemia or major hypoglycaemia
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Comb | Sita
Number analyzed (Participants) | 103 | 106
Subjects
  Target achieved | 37 | 21
  Target not achieved | 66 | 85
Statistical Analysis 1: Comparison: Comb vs Sita; Null hypothesis: Odds ratio is equal to one; Test type: Superiority or Other; p = 0.0080, Regression, Logistic — No corrections to adjust for multiplicity were performed. Statistical significance threshold was p<0.05; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.47, 95% CI [1.26 to 4.81]

4. Secondary Outcome: Number of Subjects Achieving HbA1c Less Than or Equal to 6.5%
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Comb | Sita
Number analyzed (Participants) | 103 | 106
Subjects
  Target achieved | 20 | 11
  Target not achieved | 83 | 95
Statistical Analysis 1: Comparison: Comb vs Sita; Null hypothesis: Odds ratio is equal to one; Test type: Superiority or Other; p = 0.063, Regression, Logistic — No corrections to adjust for multiplicity were performed. Statistical significance threshold was p<0.05; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.23, 95% CI [0.96 to 5.20]

5. Secondary Outcome: Number of Subjects Achieving HbA1c Less Than or Equal to 6.5% Without Symptomatic Hypoglycaemia
Description: Symptomatic hypoglycaemia is biochemically confirmed hypoglycaemia or major hypoglycaemia
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Comb | Sita
Number analyzed (Participants) | 103 | 106
Subjects
  Target achieved | 15 | 8
  Target not achieved | 88 | 98
Statistical Analysis 1: Comparison: Comb vs Sita; Null hypothesis: Odds ratio is equal to one; Test type: Superiority or Other; p = 0.135, Regression, Logistic — No corrections to adjust for multiplicity were performed. Statistical significance threshold was p<0.05; Odds Ratio (OR) = 2.07, 95% CI [0.8 to 5.37] — Treatment group comparison using logistic regression model incl.treatment,stratification factor, country as fixed effects, baseline HbA1c as covariate

6. Secondary Outcome: Change in BMI (Body Mass Index)
Time Frame: Week 0, Week 26
Population: as for outcome 2
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Comb | Sita
Number analyzed (Participants) | 103 | 107
kg/m^2 | -0.30 (0.15) | -0.58 (0.14)
Statistical Analysis 1: Comparison: Comb vs Sita; Test type: Superiority or Other; p = 0.121, ANCOVA — No corrections to adjust for multiplicity were performed. Statistical significance threshold was p<0.05; An analysis of covariance (ANCOVA) was used; baseline was included as covariate and treatment, stratification and country was included as factors; Mean Difference (Final Values) = 0.28, 95% CI [-0.07 to 0.63]

7. Secondary Outcome: Change in Body Weight
Time Frame: Week 0, Week 26
Population: as for outcome 2
Measure: Mean (Standard Error); unit: kg
Arm/Group | Comb | Sita
Number analyzed (Participants) | 103 | 107
kg | -0.81 (0.44) | -1.66 (0.42)
Statistical Analysis 1: Comparison: Comb vs Sita; Test type: Superiority or Other; p = 0.109, ANCOVA — No corrections to adjust for multiplicity were performed. Statistical significance threshold was p<0.05; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.84, 95% CI [-0.19 to 1.88]

8. Secondary Outcome: FPG (Fasting Plasma Glucose)
Time Frame: Week 26
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Comb | Sita
Number analyzed (Participants) | 103 | 106
mmol/L | 6.08 (0.24) | 8.52 (0.23)
Statistical Analysis 1: Comparison: Comb vs Sita; Test type: Superiority or Other; p = 0.0010, ANCOVA — No corrections to adjust for multiplicity were performed. Statistical significance threshold was p<0.05; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -2.45, 95% CI [-3.01 to -1.88]

9. Secondary Outcome: Hypoglycemic Episodes
Description: Overall: All episodes. Minor: Symptomatic, with PG < 3.1 mmol/L. Symptoms only: Symptomatic with PG ≥ 3.1 mmol/L
Time Frame: Weeks 0-26
Population: SAS (safety analysis set) is all randomised subjects exposed to at least one dose of trial product.
Measure: Number; unit: episodes
Arm/Group | Comb | Sita
Number analyzed (Participants) | 107 | 110
episodes
  Overall | 1 | 1
  Minor | 0 | 0
  Symptoms Only | 0 | 0
  Unclassified | 0 | 0

10. Secondary Outcome: Hypoglycemic Episodes: Day Time
Description: Day time: Episodes between 6 pm and 11 am. Overall: All episodes. Minor: Symptomatic, with PG < 3.1 mmol/L. Symptoms only: Symptomatic with PG ≥ 3.1 mmol/L
Time Frame: Weeks 0-26
Population: SAS (safety analysis set) is all randomised subjects exposed to at least one dose of trial product.
Measure: Number; unit: episodes
Arm/Group | Comb | Sita
Number analyzed (Participants) | 107 | 110
episodes
  Overall | 1 | 1
  Minor | 0 | 0
  Symptoms Only | 0 | 0
  Unclassified | 0 | 0

11. Secondary Outcome: Hypoglycemic Episodes: Night Time
Description: Night time: Episodes between 11 am and 6 pm. Overall: All episodes. Minor: Symptomatic, with PG < 3.1 mmol/L. Symptoms only: Symptomatic with PG ≥ 3.1 mmol/L
Time Frame: Weeks 0-26
Population: SAS (safety analysis set) is all randomised subjects exposed to at least one dose of trial product.
Measure: Number; unit: episodes
Arm/Group | Comb | Sita
Number analyzed (Participants) | 107 | 110
episodes
  Overall | 0 | 0
  Minor | 0 | 0
  Symptoms Only | 0 | 0
  Unclassified | 0 | 0

12. Secondary Outcome: Self-measured 9-point Plasma Glucose Profile
Time Frame: Week 26
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Comb | Sita
Number analyzed (Participants) | 98 | 98
mmol/L
  Before breakfast | 6.16 (0.20) | 8.17 (0.20)
  120 minutes after start of breakfast | 8.82 (0.28) | 10.50 (0.28)
  Before Lunch | 6.99 (0.26) | 8.01 (0.26)
  120 minutes after start of lunch | 8.69 (0.28) | 9.99 (0.28)
  Before dinner | 7.85 (0.31) | 8.61 (0.31)
  120 minutes after start of dinner | 9.30 (0.32) | 10.20 (0.32)
  Bedtime | 8.38 (0.32) | 9.42 (0.31)
  At 03:00 A.M. | 6.85 (0.26) | 8.02 (0.26)
  Before breakfast the following day | 6.07 (0.19) | 7.87 (0.19)
Statistical Analysis 1: Comparison: Comb vs Sita; Test type: Superiority or Other; Linear Mixed-model; PG profile analysis:linear mixed effect model.Treatment,time,country,time-by-treatment interaction as explanatory variables.Subject as a random factor; Mean Difference (Final Values) = -2.01, 95% CI [-2.50 to -1.51] — COMB-SITA Difference. Before breakfast
Statistical Analysis 2: Comparison: Comb vs Sita; Test type: Superiority or Other; Linear Mixed-model; [statistical method as in outcome 12, analysis 1]; Mean Difference (Final Values) = -1.64, 95% CI [-2.40 to -0.89] — COMB-SITA Difference. 120 minutes after start of breakfast
Statistical Analysis 3: Comparison: Comb vs Sita; Test type: Superiority or Other; Linear Mixed-model; [statistical method as in outcome 12, analysis 1]; Mean Difference (Final Values) = -1.02, 95% CI [-1.69 to -0.35] — COMB-SITA Difference. Before lunch
Statistical Analysis 4: Comparison: Comb vs Sita; Test type: Superiority or Other; Linear mixed-model; [statistical method as in outcome 12, analysis 1]; Mean Difference (Final Values) = -1.30, 95% CI [-2.05 to -0.56] — COMB-SITA Difference. 120 minutes after start of lunch
Statistical Analysis 5: Comparison: Comb vs Sita; Test type: Superiority or Other; Linear Mixed-model; [statistical method as in outcome 12, analysis 1]; Median Difference (Final Values) = -0.77, 95% CI [-1.58 to 0.05] — COMB-SITA Difference. Before dinner
Statistical Analysis 6: Comparison: Comb vs Sita; Test type: Superiority or Other; Linear Mixed-model; [statistical method as in outcome 12, analysis 1]; Median Difference (Final Values) = -0.88, 95% CI [-1.75 to -0.02] — COMB-SITA Difference. 120 minutes after start of dinner
Statistical Analysis 7: Comparison: Comb vs Sita; Test type: Superiority or Other; Linear Mixed-model; [statistical method as in outcome 12, analysis 1]; Mean Difference (Final Values) = -1.04, 95% CI [-1.88 to -0.20] — COMB-SITA Difference. Bedtime
Statistical Analysis 8: Comparison: Comb vs Sita; Test type: Superiority or Other; Linear Mixed Model; [statistical method as in outcome 12, analysis 1]; Mean Difference (Final Values) = -1.17, 95% CI [-1.84 to -0.49] — COMB-SITA Difference. At 03:00 a.m
Statistical Analysis 9: Comparison: Comb vs Sita; Test type: Superiority or Other; Linear Mixed-model; [statistical method as in outcome 12, analysis 1]; Mean Difference (Final Values) = -1.80, 95% CI [-2.26 to -1.34] — COMB-SITA Difference. Before breakfast the following day

ADVERSE EVENTS:
Time Frame: Weeks 0-26
Description: Safety Analysis Set is all participants treated with trial product.
Arm/Group | Comb | Sita
Serious Adverse Events (participants affected / at risk) | 2/107 | 4/110
Other Adverse Events (participants affected / at risk) | 76/107 | 72/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comb (N=107) | Sita (N=110)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Fibromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Comb (N=107) | Sita (N=110)
Nasopharyngitis (Infections and infestations) | 10/76 (13) | 14/72 (16)
Upper Respiratory Tract Infection (Infections and infestations) | 7/76 (7) | 10/72 (12)
Influenza (Blood and lymphatic system disorders) | 8/76 (9) | 4/72 (4)
Bronchitis (Blood and lymphatic system disorders) | 4/76 (4) | 4/72 (4)
Nausea (Gastrointestinal disorders) | 5/76 (7) | 8/72 (20)
Dyspepsia (Gastrointestinal disorders) | 5/76 (11) | 3/72 (11)
Headache (Nervous system disorders) | 11/76 (17) | 13/72 (32)
Dizziness (Nervous system disorders) | 3/76 (3) | 4/72 (21)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/76 (4) | 4/72 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 8/76 (9) | 2/72 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3/76 (4) | 5/72 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 4/76 (4) | 2/72 (2)
Fatigue (General disorders) | 7/76 (8) | 1/72 (1)
Asthenia (General disorders) | 0/76 (0) | 5/72 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 3/76 (3) | 5/72 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2/76 (2) | 11/72 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right not to release data before passing specified milestones. This includes the right not to release interim results that may later be found to be incorrect. At the end of the trial, one or more manuscripts will be prepared in collaboration between Investigator(s) and Novo Nordisk. Novo Nordisk will not suppress or veto publications but will reserve the right to postpone publication and/or communication for a short time to protect intellectual property.